CLINICAL TRIAL: NCT06271421
Title: Application of Nanoparticles for Cyclic Hyperthermia In Adjuvant Therapy of gLioblastoma Multiforme (ANCHIALE)
Brief Title: NanoTherm In Adjuvant Therapy of Glioblastoma Multiforme
Acronym: ANCHIALE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Collaborators: MagForce USA (Industry)
Responsible Party: Principal Investigator, Slawomir Michalak, MD, PhD, Prof., head of department, Poznan University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01/24
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Glioblastoma Multiforme
Keywords: glioblastoma; adjuvant therapy; hyperthermia; NanoTherm; GBM
MeSH Terms: conditions — Glioblastoma; Hyperthermia | interventions — Temozolomide

STUDY DESIGN:
Intervention Model Description: A prospective longitudinal study will be performed recurrent glioblastoma multiforme patients who:
  1. are included for NanoTherm therapy (group A),
  2. are included for standard Stupp protocol (surgery/chemo-radiotherapy) (group B)
Masking Description: ANCHIALE is open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NanoTherm arm (group A) (Active Comparator): Recurrent glioblastoma multiforme patients treated with NanoTherm therapy.
  Interventions: Device: NanoTherm therapy; Procedure: Glioma Resection
- Stupp protocol (group B) (Placebo Comparator): Glioblastoma multiforme patients treated according to Stupp protocol including surgery, chemotherapy and radiotherapy.
  Interventions: Procedure: Glioma Resection; Radiation: radiotherapy according to Stupp protocol; Drug: chemotherapy according to Stupp protocol

INTERVENTIONS:
Device: NanoTherm therapy — Cyclic hyperthermia in patients with recurrent glioblastoma multiforme, who underwent implantation of iron oxide nanoparticles.
  Other Names: Cyclic hyperthermia
  Arms: NanoTherm arm (group A)
Procedure: Glioma Resection — Removal of brain tumor - gross total ressection
  Other Names: Surgical removal of Glioma tumor
Radiation: radiotherapy according to Stupp protocol — The total dose according to the Stupp protocol is 60 Gy and is administered in fractions of 2 Gy per day for 5 days (Monday to Friday) for 6 weeks.
  Arms: Stupp protocol (group B)
Drug: chemotherapy according to Stupp protocol — Temozolomide is used during radiotherapy: 75 mg/m2 of body surface area per day for 7 days a week. After the completion of radiotherapy, temozolomide is used as adjuvant therapy - 6 cycles of 150-200 mg/m2 of body surface area for 5 days every 28 days.
  Other Names: temozolomide
  Arms: Stupp protocol (group B)

SUMMARY:
Glioblastoma multiforme (GBM), the most common and malignant primary brain tumor in adults is classified as a World Health Organisation (WHO) grade 4. Surgical removal of the tumor is the primary method of treatment. Unfortunately, because GBM is a disease of the entire brain, total resection is not possible. Therefore, the use of radiotherapy and/or chemotherapy is considered as Stupp protocol. Patients with recurrent GBM will be included in the ANCHIALE study.

The goal of the trial is to evaluate the efficacy and tolerance of using the NanoTherm therapy system in recurrent GBM.

The main questions it aims to answer are:

1. how NanoTherm therapy influences overall survival, and progression free survival;
2. what is the tolerance of NanoTherm therapy in terms of side effects (allergies, intracranial bleeding, infections, brain edema, increased intracranial pressure) and quality of life.

Participants will undergo:

* initial visit, considering the inclusion/exclusion criteria, neurological examination, and surveys regarding daily functioning and quality of life;
* standard neurosurgical operation aimed, if possible, complete removal of the recurrent GBM and administration of NanoTherm ASI - a sterile suspension of iron oxide nanoparticles. A catheter will be implanted allowing for measurement of temperature during the first activation in the magnetic field;
* between the 6th and 10th day after tumor resection, a standard computerized tomography (CT) scan of the head will be performed for routine postoperative evaluation;
* after the first activation (10th day), the catheter will be removed;
* subsequently, for 6 times, the patient will be subjected to the variable magnetic field of the NanoActivator® to induce hyperthermia - activations will be conducted on the 10th, 14th, 17th, 21st, 24th, and 28th day;
* for up to 2 years post-procedure, a CT scan with an evaluation of treatment efficacy will be performed;
* during follow-up visits for up to 2 years after the surgical procedure, a neurological examination, assessment of adverse symptoms, number of hospitalizations, number of medical visits, clinimetric assessment regarding quality of life, neurological deficit and degree of disability will be conducted.

Researchers will compare NanoTherm group with patients undergoing Stupp protocol treatment for the abovementioned effects.

DETAILED DESCRIPTION:
Glioblastoma multiforme (GBM) is the most frequent glial tumor (glioma). The epidemiology of brain gliomas depends on many factors such as age, gender, genetics, environment, and lifestyle.

According to statistics, in developed countries, brain gliomas account for about 2% of all tumors. In the USA, there are approximately 12,000 new cases of brain gliomas annually, and in Europe, there are about 25,000. The average age of individuals diagnosed with brain gliomas is 64 years, although they can occur in all age groups. However, the majority of cases are diagnosed in individuals between 45 and 70 years of age. The global incidence rate is 3.7/100,000 for men and 2.6/100,000 for women. A higher incidence rate is observed in highly industrialized countries. It is estimated that gliomas account for 30 to 40% of all intracranial tumors. Approximately 50% of adult gliomas are the most malignant form - Glioblastoma multiforme G4.

In 2009, 1444 new cases of malignant brain tumors were recorded in men and 1362 in women in Poland. Men have a slightly higher risk of developing brain gliomas than women. The presence of genetic and hereditary factors, including mutations in genes related to DNA repair and cell cycle control, increases the risk of developing gliomas. Risk factors for the development of gliomas include exposure to ionizing radiation and viral infections (cytomegalovirus), smoking, alcohol abuse, overweight, lack of physical activity, as well as exposure to certain chemicals such as pesticides and solvents.

Recommendations for the treatment of Glioblastoma multiforme include:

Surgical removal of the tumor as the primary method of treatment. Unfortunately, considering the fact that Glioblastoma multiforme is a disease of the entire brain, complete tumor resection is not possible. Therefore, the use of radiotherapy and/or chemotherapy is considered. This treatment is used according to the protocol published by Stupp in 2005.

Radiotherapy: Radiotherapy is used to destroy the remaining tumor cells after the tumor removal. It can be used after surgery or as a standalone treatment, especially in cases where the tumor cannot be surgically removed. The total dose according to the Stupp protocol is 60 Gy and is administered in fractions of 2 Gy per day for 5 days (Monday to Friday) for 6 weeks.

Chemotherapy: In the Stupp protocol, temozolomide is used during radiotherapy: 75 mg/m2 of body surface area per day for 7 days a week. After the completion of radiotherapy, temozolomide is used as adjuvant therapy - 6 cycles of 150-200 mg/m2 of body surface area for 5 days every 28 days.

However, the clinical effects of using the Stupp protocol are not fully satisfactory. The two-year survival rate after the full Stupp protocol (radio- and chemotherapy) is 26.5% of patients, and after using only radiotherapy, it is 10.4% of patients.

Supportive treatment methods used in the treatment of Glioblastoma multiforme so far include thermotherapy - hyperthermia and nanotherapy.

Hyperthermia involves:

* the use of elevated temperature to increase the effectiveness of radio- and chemotherapy
* thermoablation, in which the use of high temperatures - above 45°C - causes direct damage to tumor cells,
* magnetic hyperthermia (MHT), e.g. NanoTherm® Therapy (NTT), which has been registered in Europe as a method of treating Glioblastoma multiforme in cases of tumor recurrence Nanotherapy uses magnetic nanoparticles (MNP), which are used in diagnostic and therapeutic procedures.

Hyperthermia and thermotherapy have been treatment methods studied in cancer patients and magnetic hyperthermia induced using nanoparticles is becoming the subject of increasingly advanced research.

In a phase III study, the use of tumor-treating fields (TTF) was evaluated as a first-line therapy in patients with Glioblastoma multiforme. Low-power electromagnetic fields using long waves are directed at the tumor area using external electrodes. According to the report from the Institute for Quality and Efficiency in Health Care (IQWiG), this method resulted in a 5-month extension of the overall survival of patients with Glioblastoma multiforme compared to patients treated with temozolomide, and the tolerance of the treatment was acceptable.

On the other hand, NanoTherm therapy represents a promising form of thermotherapy leading to an extension of survival, especially in cases of Glioblastoma multiforme recurrence. In the study by Maier-Hauff et al., it was shown that the average overall survival of patients undergoing NanoTherm therapy after recurrence was 13.4 months, which was longer (P<0.01) than in patients treated according to the Stupp protocol (6.2 months). The overall survival after the initial diagnosis of Glioblastoma multiforme was also longer (23.2 versus 14.6 months; P<0.01). The benefit observed in both groups of patients was attributed to the use of NanoTherm therapy.

Therefore, among the sought-after new methods of treating Glioblastoma multiforme that could increase the effectiveness of the current treatment, NanoTherm therapy is a procedure that significantly increases the survival and quality of life of patients. For this reason, it is planned to conduct this study, the aim of which is to determine the effectiveness and tolerance of using nanoparticles in cyclic hyperthermia as adjuvant therapy in patients with Glioblastoma multiforme.

The main goal of the treatment for each patient with Glioblastoma multiforme is to prolong survival time and improve the quality of life. According to the literature, the median overall survival of these patients is 9 - 12 months.

Patients with recurrent glioblastoma multiforme WHO G4 will be included in the ANCHIALE study.

Study Objective:

The aim of the ANCHIALE study is to prepare a registry that allows for the evaluation of the efficacy and tolerance of using the NanoTherm therapy system in cases of recurrent glioblastoma multiforme.

Study Principles:

During the initial visit, a qualification for treatment will be conducted, taking into account the inclusion and exclusion criteria, i.e., indications and contraindications for the NanoTherm therapy system. Additionally, an interview, neurological examination, and surveys regarding daily functioning and quality of life will be conducted.

After qualifying a patient for the study, he or she will undergo standard neurosurgical operation aimed at partial or, if possible, complete removal of the recurrent brain tumor. Then, in the place of the removed tumor, NanoTherm ASI will be administered in a quantity of either 112 or 335 mg/ml of iron particles. This is a sterile suspension of iron oxide nanoparticles in sterile water, characterized by a high specific ability to absorb heat associated with its superparamagnetic properties. At the site where the thickest layer of nanoparticles (NanoTherm® ASI) is applied, a catheter will be implanted allowing for measurement and control of temperature during the first activation in the magnetic field of the NanoActivator®.

Between the 6th and 10th day after the neurosurgical procedure, a standard computerized tomography (CT) scan of the head will be performed for routine postoperative evaluation.

After the first activation (10th day post-implantation of NanoTherm® ASI), the catheter will be removed. Subsequently, cyclically, for 6 times, the patient will be subjected to the variable magnetic field of the NanoActivator® to induce hyperthermia, i.e., increase the temperature of the site after the removed tumor and the surrounding tissues. Activations will be conducted on the 10th, 14th, 17th, 21st, 24th, and 28th day. The heat released by the nanoparticles (NanoTherm® ASI) into the surrounding tissue causes destruction or damage to the cells of the glioblastoma multiforme (hyperthermia effect), increasing their susceptibility to radiotherapy and chemotherapy.

The patient will then be subjected to detailed observation for 2 years. Observation will include visits conducted on the 60th, 90th, 150th, 210th, 270th, and 360th day after surgery, and then every 3 months up to 2 years post-procedure.

On the 6th - 10th, 90th, 150th, 210th, 270th, and 360th day after surgery, and then every 3 months up to 2 years post-procedure, a CT scan with an evaluation of treatment efficacy will be performed. The treatment effects on CT will be analyzed using RANO (Response Assessment in Neuro-oncology) scale.

During follow-up visits on the 60th, 90th, 150th, 210th, 270th, and 360th day, and then every 3 months up to 2 years after the surgical procedure, a neurological examination, assessment of adverse symptoms, number of potential hospitalizations, number of medical visits, clinimetric assessment regarding quality of life (EuroQuality of Life-5 dimensions 5- levels [EQ-5D-5L], Neurologic Assessment in Neuro-Oncology [NanoScale 2]), and clinimetric assessment regarding neurological deficit and degree of disability will be conducted (modified Rankin scale, Barthel index).

The results from NanoTherm group will be compared to patients undergoing standard neurosurgical treatment for the abovementioned effects.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrence of glioblastoma multiforme.
2. Age > 18 years.
3. Informed written consent to participate in the study.
4. Karnofsky performance score ≥ 60.
5. Expected survival time > 6 months.
6. Failure of standard treatment according to the Stupp protocol.
7. Cardio-respiratory fitness - allowing to stay for 60 minutes in a lying position in the field activator.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. More than 3 foci of glioblastoma multiforme.
3. Tumor invasion of eloquent or motor areas.
4. Subependymal contrast enhancement in the adjacent brain ventricles.
5. Concurrent immunotherapy for glioblastoma.
6. Metal implants within ≤ 40 cm of the planned exposure field: metal dental fillings/restorations, cervical spine implants, metal elements left after previous craniotomies, metal elements used in osteosynthesis after orthopedically treated injuries, vascular ports with metal components.
7. Electronic implants: pacemakers, cardioverter defibrillators, cochlear implants, deep brain stimulation (DBS) electrodes.
8. Allergy/hypersensitivity to aminosilanes, iron oxide, acetic acid.
9. Planned or current treatment with electromagnetic field in the Optune®TTF system.
10. Claustrophobia not amenable to control.
11. Painful conditions, musculoskeletal system diseases that prevent staying in a lying position.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Survival following the surgery [units months 1-24] | 2 years following surgery
  overall survival
Progression free survival [units months 1-24] | 2 years after surgery
  Progression Free Survival

SECONDARY OUTCOMES:
Response Assessment in Neuro-oncology [1 - complete response; 4 -progressive disease] | 2 years after surgery
  Response Assessment in Neuro-oncology - the scale describes the response to the treatment basing on neuroimaging.
EuroQuality of Life 5-dimensions-5 levels scale (EQ-5D-5L) [arbitraty units 0- worst ; 100 - best] | 2 years after surgery
  quality of life - This scale is numbered from 0 to 100; 100 means the best health you can imagine; 0 means the worst health you can imagine.
Neurologic Assessment in Neuro-Oncology (NanoScale 2) [0-best; 23-worst] | 2 years after surgery
  functional assessment of the nervous system: 0 - no deficit, 23 - severe neurological deficit
modified Rankin scale [0-best; 6-worst] | 2 years after surgery
  disability scale
Barthel index [range 0-100; 0-best, 100-worst] | 2 years after surgery
  measure of performance in activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Slawomir Michalak, Prof., Principal Investigator — Poznan University of Medical Sciences
Locations (1):
- University Hospital, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Barker CA, Chang M, Chou JF, Zhang Z, Beal K, Gutin PH, Iwamoto FM. Radiotherapy and concomitant temozolomide may improve survival of elderly patients with glioblastoma. J Neurooncol. 2012 Sep;109(2):391-7. doi: 10.1007/s11060-012-0906-4. Epub 2012 Jun 12. PMID 22688802
- [Background] Gupta T, Sarin R. Poor-prognosis high-grade gliomas: evolving an evidence-based standard of care. Lancet Oncol. 2002 Sep;3(9):557-64. doi: 10.1016/s1470-2045(02)00853-7. PMID 12217793
- [Background] Sun J, Guo M, Pang H, Qi J, Zhang J, Ge Y. Treatment of malignant glioma using hyperthermia. Neural Regen Res. 2013 Oct 15;8(29):2775-82. doi: 10.3969/j.issn.1673-5374.2013.29.009. PMID 25206588
- [Background] Mahmoudi K, Bouras A, Bozec D, Ivkov R, Hadjipanayis C. Magnetic hyperthermia therapy for the treatment of glioblastoma: a review of the therapy's history, efficacy and application in humans. Int J Hyperthermia. 2018 Dec;34(8):1316-1328. doi: 10.1080/02656736.2018.1430867. Epub 2018 Feb 6. PMID 29353516
- [Background] Maier-Hauff K, Ulrich F, Nestler D, Niehoff H, Wust P, Thiesen B, Orawa H, Budach V, Jordan A. Efficacy and safety of intratumoral thermotherapy using magnetic iron-oxide nanoparticles combined with external beam radiotherapy on patients with recurrent glioblastoma multiforme. J Neurooncol. 2011 Jun;103(2):317-24. doi: 10.1007/s11060-010-0389-0. Epub 2010 Sep 16. PMID 20845061
- [Background] Pinel S, Thomas N, Boura C, Barberi-Heyob M. Approaches to physical stimulation of metallic nanoparticles for glioblastoma treatment. Adv Drug Deliv Rev. 2019 Jan 1;138:344-357. doi: 10.1016/j.addr.2018.10.013. Epub 2018 Nov 7. PMID 30414495
- [Background] Boroon MP, Ayani MB, Bazaz SR. Estimation of the optimum number and location of nanoparticle injections and the specific loss power for ideal hyperthermia. J Therm Biol. 2018 Feb;72:127-136. doi: 10.1016/j.jtherbio.2018.01.010. Epub 2018 Jan 31. PMID 29496005
- [Background] Grauer O, Jaber M, Hess K, Weckesser M, Schwindt W, Maring S, Wolfer J, Stummer W. Combined intracavitary thermotherapy with iron oxide nanoparticles and radiotherapy as local treatment modality in recurrent glioblastoma patients. J Neurooncol. 2019 Jan;141(1):83-94. doi: 10.1007/s11060-018-03005-x. Epub 2018 Dec 1. PMID 30506500
- [Background] Huang H, Yu K, Mohammadi A, Karanthanasis E, Godley A, Yu JS. It's Getting Hot in Here: Targeting Cancer Stem-like Cells with Hyperthermia. J Stem Cell Transplant Biol. 2017;2(2):113. Epub 2017 Dec 29. PMID 30542674
- [Background] Curran WJ Jr, Scott CB, Horton J, Nelson JS, Weinstein AS, Fischbach AJ, Chang CH, Rotman M, Asbell SO, Krisch RE, et al. Recursive partitioning analysis of prognostic factors in three Radiation Therapy Oncology Group malignant glioma trials. J Natl Cancer Inst. 1993 May 5;85(9):704-10. doi: 10.1093/jnci/85.9.704. PMID 8478956
- [Background] Dong X, Noorbakhsh A, Hirshman BR, Zhou T, Tang JA, Chang DC, Carter BS, Chen CC. Survival trends of grade I, II, and III astrocytoma patients and associated clinical practice patterns between 1999 and 2010: A SEER-based analysis. Neurooncol Pract. 2016 Mar;3(1):29-38. doi: 10.1093/nop/npv016. Epub 2015 Jul 1. PMID 31579519
- [Background] Gupta R, Sharma D. Evolution of Magnetic Hyperthermia for Glioblastoma Multiforme Therapy. ACS Chem Neurosci. 2019 Mar 20;10(3):1157-1172. doi: 10.1021/acschemneuro.8b00652. Epub 2019 Feb 19. PMID 30715851
- [Background] Hegi ME, Liu L, Herman JG, Stupp R, Wick W, Weller M, Mehta MP, Gilbert MR. Correlation of O6-methylguanine methyltransferase (MGMT) promoter methylation with clinical outcomes in glioblastoma and clinical strategies to modulate MGMT activity. J Clin Oncol. 2008 Sep 1;26(25):4189-99. doi: 10.1200/JCO.2007.11.5964. PMID 18757334
- [Background] Laperriere N, Zuraw L, Cairncross G; Cancer Care Ontario Practice Guidelines Initiative Neuro-Oncology Disease Site Group. Radiotherapy for newly diagnosed malignant glioma in adults: a systematic review. Radiother Oncol. 2002 Sep;64(3):259-73. doi: 10.1016/s0167-8140(02)00078-6. PMID 12242114
- [Background] Nwokedi EC, DiBiase SJ, Jabbour S, Herman J, Amin P, Chin LS. Gamma knife stereotactic radiosurgery for patients with glioblastoma multiforme. Neurosurgery. 2002 Jan;50(1):41-6; discussion 46-7. doi: 10.1097/00006123-200201000-00009. PMID 11844233
- [Background] Paszat L, Laperriere N, Groome P, Schulze K, Mackillop W, Holowaty E. A population-based study of glioblastoma multiforme. Int J Radiat Oncol Biol Phys. 2001 Sep 1;51(1):100-7. doi: 10.1016/s0360-3016(01)01572-3. PMID 11516858
- [Background] Stupp R, Taillibert S, Kanner A, Read W, Steinberg D, Lhermitte B, Toms S, Idbaih A, Ahluwalia MS, Fink K, Di Meco F, Lieberman F, Zhu JJ, Stragliotto G, Tran D, Brem S, Hottinger A, Kirson ED, Lavy-Shahaf G, Weinberg U, Kim CY, Paek SH, Nicholas G, Bruna J, Hirte H, Weller M, Palti Y, Hegi ME, Ram Z. Effect of Tumor-Treating Fields Plus Maintenance Temozolomide vs Maintenance Temozolomide Alone on Survival in Patients With Glioblastoma: A Randomized Clinical Trial. JAMA. 2017 Dec 19;318(23):2306-2316. doi: 10.1001/jama.2017.18718. PMID 29260225
- See also: IQWiG, Institut für Qualität und Wirtschaftlichkeit im Gesundheitswesen, 2019. — https://www.iqwig.de/download/n18-02_tumortherapiefelder-beim-glioblastom_rapid-report_v1-1.pdf?rev=186827
- See also: Tadashi Osawa et al. Elderly patients aged over 75 years with glioblastoma: Preoperative status and surgical strategies. — https://doi.org/10.1016/j.inat.2021.101127